CLINICAL TRIAL: NCT02783937
Title: Filgrastim for Treatment of Premature Ovarian Insufficiency: Randomized Clinical Trial
Brief Title: Filgrastim for Premature Ovarian Insufficiency
Acronym: FIL-POI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammad Abdel-Rahman Mohammad Ahmed, Doctor, South Valley University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OBGYN001
Record Dates: First submitted 2016-05-17; First posted 2016-05-26 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Premature Ovarian Failure
Keywords: Premature; Ovarian; Failure; Filgrastim
MeSH Terms: conditions — Primary Ovarian Insufficiency; Premature Birth | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filgrastim arm (Active Comparator): Intervention: Filgrastim vial (30 million IU/ml) SC injection twice daily for five consecutive days
  Interventions: Biological: Filgrastim
- Placebo arm (Placebo Comparator): Intervention: Injection of saline SC injection twice daily for five consecutive days.
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Filgrastim — Each case will have two intervention phases done blindly at random with a wash-out period of 6 months:
  Phase A:
  Filgrastim vial (30 million IU/ml) SC injection twice daily for five consecutive days.
  Phase B:
  Injection of saline SC injection twice daily for five consecutive days.
  Other Names: Granulocyte-Colony Stimulating Factor (G-CSF)
  Arms: Filgrastim arm
Drug: Saline — Injection of saline SC injection twice daily for five consecutive days
  Other Names: placebo
  Arms: Placebo arm

SUMMARY:
Filgrastim is a Granulocyte-Colony Stimulating factor (G-CSF). It is an FDA approved drug. Very small embryonic-like stem cells (VSELs) are found in the ovary. Animal studies showed that these cells are able to regenerate the affected ovary. Studies on mice have shown that Filgrastim result in recovery of oogenesis after chemotherapy-induced gonadal failure (in 2013, 2014, and 2015).

DETAILED DESCRIPTION:
Premature ovarian insufficiency (POI) has no curative treatment until now. Filgrastim is an FDA approved Granulocyte-Colony Stimulating factor (G-CSF). Very small embryonic-like stem cells (VSELs) are found in the testis and ovary. VSELs are stem cells that have noticed to survive chemotherapy induced gonadal failure. Data from animal studies showed that stimulation of these stem cells result in generation of the affected gonads. Studies on mice have shown a promising stimulating effect of Filgrastim on recovery of spermatogenesis and oogenesis after chemotherapy-induced gonadal failure (in 2013, 2014, and 2015).

ELIGIBILITY:
Inclusion Criteria:

* Women with Premature Ovarian Insufficiency (POI): For the purpose of the research women is considered to have POI if she is aged less than 40 years and has amenorrhea of at least 4 month with FSH level above 25 IU/L (repeated twice >4 weeks apart).

Exclusion Criteria:

* Abnormal karyotype
* Previous pelvic or abdominal radiotherapy
* Previous surgical removal of the ovarian pathology
* Chronic disease: renal, liver, cardiac, malignancy

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11; Primary Completion 2020-12 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Return of menses | 6 months
  Return of menses in patients with amenorrhea of at least 4 months

SECONDARY OUTCOMES:
Pregnancy | 6 months
  Occurrence of pregnancy as diagnosed by positive serum B-hCG and/or ultrasound
serum Estradiol | 6 months
  Normalization of serum Estradiol as tested bi-weekly
serum Anti-mullarian Hormone (AMH) | 6 months
  Normalization of serum AMH in patients with AMH level less than 0.9 ng/mL
serum FSH | 6 months
  Normalization of serum FSH in patients with FSH level above 25 IU/L
Follicular growth | 6 months
  Growth of follicle to size at least 18 mm as monitored by transvaginal ultrasound
endometrial thickness | 6 months
  increase of endometrial thickness in women with thin endometrium (less then 8 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad AM Ahmed, MD, Principal Investigator — Egypt, Qena, South Valley University, faculty of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skaznik-Wikiel ME, McGuire MM, Sukhwani M, Donohue J, Chu T, Krivak TC, Rajkovic A, Orwig KE. Granulocyte colony-stimulating factor with or without stem cell factor extends time to premature ovarian insufficiency in female mice treated with alkylating chemotherapy. Fertil Steril. 2013 Jun;99(7):2045-54.e3. doi: 10.1016/j.fertnstert.2013.01.135. Epub 2013 Feb 26. PMID 23453120
- [Background] Akdemir A, Zeybek B, Akman L, Ergenoglu AM, Yeniel AO, Erbas O, Yavasoglu A, Terek MC, Taskiran D. Granulocyte-colony stimulating factor decreases the extent of ovarian damage caused by cisplatin in an experimental rat model. J Gynecol Oncol. 2014 Oct;25(4):328-33. doi: 10.3802/jgo.2014.25.4.328. Epub 2014 Jun 18. PMID 25142624
- [Background] Benavides-Garcia R, Joachim R, Pina NA, Mutoji KN, Reilly MA, Hermann BP. Granulocyte colony-stimulating factor prevents loss of spermatogenesis after sterilizing busulfan chemotherapy. Fertil Steril. 2015 Jan;103(1):270-80.e8. doi: 10.1016/j.fertnstert.2014.09.023. Epub 2014 Nov 5. PMID 25439845
- [Background] Bhartiya D, Anand S, Parte S. VSELs may obviate cryobanking of gonadal tissue in cancer patients for fertility preservation. J Ovarian Res. 2015 Nov 17;8:75. doi: 10.1186/s13048-015-0199-2. PMID 26576728
- [Background] Roness H, Kalich-Philosoph L, Meirow D. Prevention of chemotherapy-induced ovarian damage: possible roles for hormonal and non-hormonal attenuating agents. Hum Reprod Update. 2014 Sep-Oct;20(5):759-74. doi: 10.1093/humupd/dmu019. Epub 2014 May 15. PMID 24833728